CLINICAL TRIAL: NCT07390227
Title: Virtual Reality Intervention in Patients With Persistent Shoulder Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HAN University of Applied Sciences (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, Beate Dejaco, Principal Investigator at department Key Factors in Physical Activity and Rehabilitation Care, HAN University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECO 721.11/25
Record Dates: First submitted 2026-01-02; First posted 2026-02-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Rotator Cuff Syndrome; Shoulder Instability; Frozen Shoulder
Keywords: Virtual reality; Shoulder; persitent shoulder pain
MeSH Terms: conditions — Bursitis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR intervention arm (Experimental): the intervention consists of educational video's, a simulation debriefing and VR exercises at home.
  Interventions: Other: Exercise with Virtual reality; Other: education on shoulder pain; Other: simulation de-briefing

INTERVENTIONS:
Other: Exercise with Virtual reality — Participants exercise their shoulder at home with a VR headset, provided by the research team. The physiotherapist explains how to use the headset and wich applicatiosn should be used at which level. participants exercise daily 10 minutes for six weeks.
Other: education on shoulder pain — participants receive a video-clip of 3 minutes that explains their shoulder condition.
Other: simulation de-briefing — During the physiotherapy conultation, participants will be video-recorded with their own mobile device, when moving within VR. After thtat, the phyiotherapist and participant engage in a simulation de-briefing, discussing how it felt to move within VR, any changes in perceptions on pain and movement are discussed as well as the transfer to other movements in daily life.

SUMMARY:
Shoulder pain is very common and can make daily activities difficult. Many people have shoulder pain for a long time, even after treatment. Common shoulder problems include pain from the shoulder muscles and tendons, a frozen shoulder, or an unstable shoulder. Unfortunately, both surgery and physiotherapy often help only a little. This can be due to many reasons, such as people not continuing their exercises, fear of moving the shoulder, incorrect beliefs about pain, other health problems, or lifestyle factors.

Virtual Reality (VR) is a new and promising technology that is already being used to help people with long-lasting pain. By using a VR headset, people can exercise in a motivating and engaging virtual environment. VR may help reduce fear of movement, improve how people feel about their body, make movement easier, and help people stick to their exercises. However, there is still very little research on using VR for long-lasting shoulder pain.

The goal of this study is to find out whether a home-based VR exercise program for people with ongoing shoulder complaints is practical and acceptable. The investigators want to know if people are willing and able to use VR at home, whether they continue the treatment, and whether it shows early signs of reducing pain and limitations. They also want to understand who benefits most from VR, in which situations it works best, and why it may or may not help.

People aged 16 years and older who have had shoulder pain and limitations for more than three months can take part. This includes people with shoulder tendon-related pain, frozen shoulder, or shoulder instability.

The study lasts six weeks and includes three parts. First, participants receive online educational videos about shoulder pain and movement. Second, they take part in three physiotherapy sessions: one in person and two online. Third, participants use a VR headset at home every day for about 15 minutes to perform guided shoulder and whole-body exercises, such as reaching or aiming tasks. The exercises gradually become more challenging. Participants receive clear written and video instructions, and technical support is available if needed.

During the study, participants will complete questionnaires and the VR system will record basic usage data. At the end of the study, group interviews will be held with participants and physiotherapists to talk about their experiences with VR and how it influenced pain, movement, and daily activities.

Using VR is considered safe. Some people may experience mild and short-lasting side effects, such as dizziness, but serious problems are not expected. The main effort for participants is the time spent on exercises and completing questionnaires.

The results of this study will help determine whether VR is a useful and realistic treatment option for people with long-lasting shoulder pain and will guide future, larger studies.

DETAILED DESCRIPTION:
For many people the long-term disability associated with musculoskeletal disorders (MSK) is substantial. Within this group of conditions, musculoskeletal shoulder problems are ubiquitous. They impact on sleep, social interaction, ability to perform activities of daily living, sporting participation, and work. The prevalence of MSK shoulder disorders is reported to range from 0.7% to 55.2%, with the incidence ranging from 7.7 to 62.0 per thousand people per year. For people older than 65 years of age, more than 30 per cent experience shoulder pain and disability daily. These shoulder complaints encompass among others rotator cuff related shoulder pain (RCRSP), instability of the glenohumeral joint and frozen shoulders. Pharmacological, surgical, and non-surgical interventions are used in the management of persistent shoulder pain conditions, however, all current interventions for persistent shoulder conditions are associated with, at best, modest clinical effects. This limited efficacy may be attributed to several factors such as poor engagement and adherence to exercise and advice, unhelpful sickness beliefs ("the tendons will snap if I elevate the arm") and unhelpful coping strategies (fear of movement, protective movements, catastrophic thinking). These limitations highlight the need for novel, comprehensive treatment approaches that address both the physical and psychological aspects of persistent shoulder pain while promoting patient engagement and adherence.

Extended reality (XR) is an existing technology that is being increasingly integrated for use in healthcare. XR is being used for patient education, various physical, and psychological conditions, as well as pain conditions. It is being used in the management of anxiety disorders, posttraumatic stress disorders, cardiorespiratory disease, neurological disorders, and musculoskeletal conditions. Initially used in the gaming industry, different XR technologies have been rapidly introduced in various areas of healthcare. XR, which encompasses a continuum of realities such as Augmented Reality (AR), Mixed Reality (MR), and Immersive Virtual Reality (iVR) represents different forms of the technology. While AR and MR maintain a connection to the real world by overlaying or integrating virtual elements, immersive VR creates a fully immersive digital environment that replaces the real-world with an illusionary digital world, typically introduced within head-mounted-displays (HMDs).

XR has been shown to be effective in acute and persistent pain conditions such as painful medical procedures and wound care, knee and hip osteoarthritis, persistent low back pain, and shoulder pain. The mechanisms by which XR and especially iVR may decrease pain and disability are not fully elucidated but may be due to distraction and attentional shifting, manipulation of sensory input through multisensory feedback and embodiment that potentially alters body perception. Virtual environments encourage movement by allowing patients to move without being cognizant of how they move, how far they move, the complexity of movement, or the speed at which they move. This may enhance new movement strategies and encourage the restoration of normal movements (less guarded or protective movement). By violating negative expectations of movement34 and decreasing fear of movement, range of motion and function may be improved, and pain levels may decrease. Furthermore, VR has been reported to be engaging, enjoyable, and associated with positive feelings allowing for an increase in participation and adherence to exercise therapy.

Despite the growing interest in iVR for musculoskeletal rehabilitation, there is a notable gap in the literature regarding its application and effectiveness specifically for persistent shoulder pain. Given the evolving nature and contextual sensitivity of virtual reality (VR) interventions, this study follows the recommendation by Birckhead et al, who argue for a hypothesis-generating and exploratory approach in early-stage VR research, rather than premature large-scale randomized trials. VR is a complex, multicomponent intervention whose effectiveness likely depends on interactions between individual characteristics, contextual factors, and specific features of the technology. A purely quantitative approach might not be able to elucidate the complexities of how and why it may (or may not) work for different patients. The investigators will therefore perform a mixed-methods feasibility design, in which quantitative assessment focusing on Bowen's feasibility areas acceptability, demand, and preliminary efficacy is combined with Realist evaluation. The Realist evaluation is a theory-driven approach that seeks to understand not only whether an intervention works, but for whom, under what circumstances, and through which mechanisms. An initial initial program theory will be developped based on literature and expert input, expressed as context-mechanism-outcome configurations. The theory will then be tested through qualitative realist interviews. This allows for generating a program theory for the VR intervention and will inform both the refinement of the intervention and the design of future confirmatory trials, aligned with the UK Medical Research Council (MRC) Framework for Complex Interventions.

2. OBJECTIVES

Primary Objective:

To evaluate the feasibility in terms of acceptability, demand, and preliminary efficacy of a six-week homebased iVR intervention in patients with persistent shoulder complaints.

The recommendations for the design of a feasibility study of Bowen et al will be followed, exploring the following areas of focus of feasibility: 1) acceptability, 2) demand and 3) preliminary efficacy.

1) Focus area acceptability:

1. recruitment rate defined as the number of participants who give their consent to the orthopaedic surgeon for an appointment with the research team to screen for eligibility
2. participation rate defined as the number of participants enrolled in the study divided by the number of eligible individuals approached
3. drop-out rate defined as the proportion of participants who discontinue the study before completing the 6-week VR program

3. rate of response to questionnaires defined as the number of fully completed questionnaires at baseline and follow-up 4. usability and acceptance of the iVR intervention using the Virtual Reality System Usability Questionnaire

2) Focus area of demand:

1. adherence to study protocol by physiotherapists and patients: data collection via system logs of VR headsets (frequency of use, total time spent in VR) and data collected in focus group interviews.

3) Focus area of preliminary efficacy:

1. Pain: (NRS 0-10) for pain during the last 24h, pain at rest and pain at night
2. Disability: Shoulder Pain and Disability Index (SPADI)
3. Fear of movement: Tampa Scale for Kinesiophobia (TSK -11)
4. Illness perceptions: Brief Illness Perception Questionnaire (B-IPQ),
5. Sleep quality: Sleep Quality Scale (SQS).

Secondary Objective(s):

To explore the perceived underlying mechanisms of VR outcomes by developing an initial program theory (CMO's) and refine the initial theory through collecting data by means of focus group interviews of participating physiotherapists and patients.

Explored items will be:

* To assess how different contexts (patient, physiotherapist, and environmental factors) influence the acceptability, demand, and efficacy of the VR intervention.
* To explore the mechanisms by which immersive VR may (or may not) lead to reductions in pain, disability, fear of movement, or poor sleep.
* To identify patterns of outcomes across subgroups of patients and contexts, thereby refining the initial program theory of how VR works for persistent shoulder complaints.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria:

  * Unilateral shoulder pain NPRS ≥ 4/10, persisting longer than 3 months
  * Adults ≥ 16 years old
  * Willing and able to comply with study protocol
  * Diagnosis of rotator cuff related shoulder pain, or shoulder instability, or frozen shoulder, confirmed according to international clinical guidelines

    1. RC related shoulder pain
  * shoulder pain and/or weakness during active or resisted shoulder external rotation, and or, shoulder elevation and/or
  * Presence of Painful arc during elevation

    2. shoulder instability
  * Radiographically, computed tomography scans, magnetic resonance imaging scans confirmed dislocation or
  * Documented history of manual or surgical relocation of the shoulder
  * Traumatic onset with persistent symptoms
  * Positive apprehension sign (fear of imminent dislocation when the arm is placed in abduction and external rotation during clinical examination)

    3. frozen shoulder
  * Restricted active and passive range of shoulder movement in all directions
  * Restricted active and passive shoulder external rotation of 50 percent compared to non-painful arm
  * Nothing abnormal detected on radiograph of shoulder

Exclusion Criteria:

* Neurological disease affecting the shoulder
* Shoulder stiffness not consistent to frozen shoulder
* Pain in the shoulder that is elicited by movements of the head and neck.
* history of motion-sickness
* history of seizures
* severe vertigo or vestibular impairment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The outcome measure belongs to the following areas of focus of feasibility 1) acceptability | From enrollment to the end of the treament 7 weeks
  acceptability:
  1. recruitment rate defined as the number of participants who give their consent to the orthopaedic surgeon for an appointment with the research team to screen for eligibility
  2. participation rate defined as the number of participants enrolled in the study divided by the number of eligible individuals approached
  3. drop-out rate defined as the proportion of participants who discontinue the study before completing the 6-week VR program
  3. rate of response to questionnaires defined as the number of fully completed questionnaires at baseline and follow-up

OTHER OUTCOMES:
Focus area of demand: adherence | 7 weeks
  adherence to study protocol by physiotherapists and patients: data collection via system logs of VR headsets (frequency of use, total time spent in VR) and data collected in focus group interviews.
Focus area of preliminary efficacy: pain | 8 weeks
  Pain: (NRS 0-10) for pain during the last 24h, pain at rest and pain at night
Focus area of preliminary efficacy: | 8 weeks
  Disability: Shoulder Pain and Disability Index (SPADI)
Focus area of preliminary efficacy | 8 weeks
  Fear of movement: Tampa Scale for Kinesiophobia (TSK -11)
Focus area of preliminary efficacy | 8 weeks
  Illness perceptions: Brief Illness Perception Questionnaire (B-IPQ)
Focus area of preliminary efficacy | 8 weeks
  Sleep quality: Sleep Quality Scale (SQS).

CONTACTS AND LOCATIONS:
Overall Officials: Bart Staal, PhD, Study Director — HAN University of Applied Sciences
Locations (1):
- HAN, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Subjects will be coded by a numeric code to create an anonymous dataset. Investigators have access to this code and will store the subject identification code list at a separate location from the dataset. Data will be stored at the Radboud Data repository in accordance with the General Data Protection Regulation (in Dutch: Algemene Verordening Gegevensbescherming) and will be available on the following DOI:10.34973/xd0v-9620, after publication of the manuscript.
Supporting Information: SAP, CSR
Time Frame: after completion of the study
Access Criteria: IPD are available at the previous mentioned DOI at the Radboud Data Repository. Data From the qualitative part of the study will only have restricted access.
URL: https://dmp.radboudumc.nl/plans/87426/edit?phase_id=8714

REFERENCES:
- [Result] Rossettini G, Colombi A, Carlino E, Manoni M, Mirandola M, Polli A, Camerone EM, Testa M. Unraveling Negative Expectations and Nocebo-Related Effects in Musculoskeletal Pain. Front Psychol. 2022 Mar 16;13:789377. doi: 10.3389/fpsyg.2022.789377. eCollection 2022. PMID 35369173
- [Result] Matamala-Gomez M, Diaz Gonzalez AM, Slater M, Sanchez-Vives MV. Decreasing Pain Ratings in Chronic Arm Pain Through Changing a Virtual Body: Different Strategies for Different Pain Types. J Pain. 2019 Jun;20(6):685-697. doi: 10.1016/j.jpain.2018.12.001. Epub 2018 Dec 16. PMID 30562584
- [Result] de Vries FS, van Dongen RTM, Bertens D. Pain education and pain management skills in virtual reality in the treatment of chronic low back pain: A multiple baseline single-case experimental design. Behav Res Ther. 2023 Mar;162:104257. doi: 10.1016/j.brat.2023.104257. Epub 2023 Jan 18. PMID 36731183
- [Result] Alvarez de la Campa Crespo M, Donegan T, Amestoy-Alonso B, Just A, Combalia A, Sanchez-Vives MV. Virtual embodiment for improving range of motion in patients with movement-related shoulder pain: an experimental study. J Orthop Surg Res. 2023 Sep 26;18(1):729. doi: 10.1186/s13018-023-04158-w. PMID 37752613
- [Result] Caneiro JP, Smith A, Bunzli S, Linton S, Moseley GL, O'Sullivan P. From Fear to Safety: A Roadmap to Recovery From Musculoskeletal Pain. Phys Ther. 2022 Feb 1;102(2):pzab271. doi: 10.1093/ptj/pzab271. PMID 34971393
- [Result] Clausen MB, Merrild MB, Holm K, Pedersen MW, Andersen LL, Zebis MK, Jakobsen TL, Thorborg K. Less than half of patients in secondary care adheres to clinical guidelines for subacromial pain syndrome and have acceptable symptoms after treatment: A Danish nationwide cohort study of 3306 patients. Musculoskelet Sci Pract. 2021 Apr;52:102322. doi: 10.1016/j.msksp.2021.102322. Epub 2021 Jan 12. PMID 33485212
- [Result] Page MJ, Green S, McBain B, Surace SJ, Deitch J, Lyttle N, Mrocki MA, Buchbinder R. Manual therapy and exercise for rotator cuff disease. Cochrane Database Syst Rev. 2016 Jun 10;2016(6):CD012224. doi: 10.1002/14651858.CD012224. PMID 27283590
- [Result] GBD 2016 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2017 Sep 16;390(10100):1211-1259. doi: 10.1016/S0140-6736(17)32154-2. PMID 28919117
- See also: this page describes the whole research project on VR in shoulder rehabilitation — https://www.nwo.nl/projecten/023022010